CLINICAL TRIAL: NCT06800937
Title: Evaluation of the Sphingolipidomic Profile in Women Suffering From Anorexia Nervosa: Relationship With Clinical-endocrine and Psychiatric Parameters
Brief Title: Sphingolipidomic Profile in Anorexia Nervosa
Acronym: SFINGOANNER
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C417
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Sphingolipids; Females; Lipidomic profile
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anorexia Nervosa: Adult female Anorexia Nervosa patients, hospitalized at the Division of Eating and Nutrition Disorders (END), Istituto Auxologico Italiano, IRCCS, Piancavallo (VB), Italy
  Interventions: Other: Determination of sphingolipidomic profile
- Normal weight: Adult normal-weight women with a Body Mass Index between 18.5 and 24.9 kg/m2, recruited from research and hospital staff
  Interventions: Other: Determination of sphingolipidomic profile

INTERVENTIONS:
Other: Determination of sphingolipidomic profile — The plasma/serum levels of the following sphingolipids will be measured: ceramides and dihydroceramides from C16 to C24, including 2 unsaturated ones (C18:1 and C24:1), sphingomyelins (those from C16 to C24 and the one C24:1), sphingosine, sphinganine, sphingosine-1-phosphate and sphinganine-1-phosphate.

SUMMARY:
: The objective of this research project will be to determine the sphingolipidomic profile in a group of women (> 18 years) affected by Anorexia Nervosa (AN), phenotypically characterized (restricting [AN-R] vs binge-eating purging [AN-BP]). Specific questionnaires will be administered for the definition of the severity of the eating disorder and depressive state (suicidality), to which will be added the evaluation of gonadal function (i.e., plasma levels of estradiol/progesterone and use of oral contraceptives).

Based on the specific lipidomic profile, which the present research project hopes to characterize, it will be possible to appropriately modify the diet of rehabilitation programs and, in the future, improve the effectiveness of the treatment itself, especially in the long term.

ELIGIBILITY:
Patients with Anorexia Nervosa:

Inclusion Criteria:

* Female sex
* Age: 18 years or older
* Diagnosis of Anorexia Nervosa in the acute phase
* Hospitalized at the Division of Eating and Nutrition Disorders (END), San Giuseppe Hospital, Istituto Auxologico Italiano, IRCCS, Piancavallo (VB), Italy

Exclusion Criteria:

* Absence of signed Informed Consent

Control group:

Inclusion Criteria:

* Female sex
* Age: 18 years or older
* BMI between 18.5 and 24.9 kg/m2

Exclusion Criteria:

* Absence of signed Informed Consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 female adults with Anorexia nervosa, according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), hospitalized at the Division of Eating and Nutrition Disorders (END), San Giuseppe Hospital, Istituto Auxologico Italiano, IRCCS, Piancavallo, Italy.
  Half will have the AN-R subtype and the other AN-BP.
  30 normal weight adult women recruited from research and hospital staff, with Body Mass Index between 18.5 and 24.9 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Ceramides | Baseline
  Plasma level of ceramide
Dihydroceramides | Baseline
  Plasma level of dihydroceramides

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy